CLINICAL TRIAL: NCT05421793
Title: Towards a Food Ingredient Clinically Proven to Benefit Gut Health: Novel RG-I Variants
Brief Title: Prebiotic and Anti-inflammatory Effects of a Pectin Polysaccharide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: NutriLeads B.V. (Wageningen, The Netherlands) (Unknown)
Responsible Party: Principal Investigator, Robert Brummer, Professor, Örebro University, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-01814-02
Record Dates: First submitted 2022-06-07; First posted 2022-06-16 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: paracellular permeability; transcellular permability; rhamnogalacturonan I; prebiotic; gut microbiota

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gut barrier function treatments (Experimental): Stressor, fibre, combination of treatments.
  Interventions: Other: Fermented product of carrot derived rhamnogalacturonan I

INTERVENTIONS:
Other: Fermented product of carrot derived rhamnogalacturonan I — Stimulation of human colonic biopsies with the fermented product of carrot derived rhamnogalacturonan I

SUMMARY:
The aim of this study is to determine, quantify and understand the potential prebiotic and anti-inflammatory effects of the pecticpolysaccharide rhamnogalacturonan I (RG-I). The effects of these dietary fibre fractions on barrier function will also be investigated.

DETAILED DESCRIPTION:
The dietary fibre fractions from RG-I will be tested first for their prebiotic potential. Batch culture fermentation systems containing basal growth medium will be inoculated with faecal homogenates obtained from different time points (Task I) and will be used for analyzing microbiota composition and microbiota-associated metabolites. Subsequently, the collection of colon biopsies through sigmoidoscopy procedure of the same subjects will take place and the collected biopsies will be mounted in Ussing Chambers. Supernatants collected from Task I will be added to the mucosal side of the biopsy together with a stressor and two permeability markers, in order to investigate the effects of the fibre fractions on both paracellular and transcellular permeability.Throughout the study subjects will complete questionnaires related to their gastrointestinal health and dietary habits

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent prior to any study related procedures
2. Age 18-65 years
3. Willing to abstain from regular consumption of prebiotics/probiotics products or medication known to alter gastrointestinal functions at least 4 weeks prior to the study visits

Exclusion Criteria:

1. Previous complicated gastrointestinal surgery
2. Presence of gastrointestinal disorder or any disorder which the principal investigator considers to affect the results of the study
3. Current diagnosis of psychiatric disease
4. Current and past diagnosis inflammatory gastrointestinal disease (e.g. Irritable Bowel Disease)
5. Systemic use of antibiotics or steroids medications in the last 3 months
6. Frequent use of NSAID (Non Steroidal Anti Inflammatory Drugs) the last 2 months prior to study visits
7. Regular consumption of prebiotic/probiotic products for the past 4 weeks
8. Abuse of alcohol or drugs
9. Frequent use of laxatives, anti-diarrheal, anti-cholinergic within last 12 weeks prior to study visits
10. Pregnancy and breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of barrier function after 90 minutes of ex vivo stimulation of the colonic biopsies. | Barrier function will be measured at baseline and after 90 minutes of ex vivo stimulation of the colonic biopsies.
  Barrier function will be evaluated with the use of markers related to paracellular and transcellular permeability, through immunofluoresence and ELISA tecnhique.
Change from baseline to the effect on the intestinal microbial populations and their metabolic products [i.e. Short-Chain Fatty Acids (SCFA)] (prebiotic effect) by the end of the in vitro fermentation process. | The levels of microbial populations and their metabolic products will be measured at baseline and after 6 hours of in vitro fermentation procedure.
  Microbial populations will be quantified with 16SRNA sequencing and quantitative Polymerase Chain Reaction (PCR).
  SCFAs will be quantified with Gas chromatography.

SECONDARY OUTCOMES:
Effect of RG-I fractions on immune system reinforcement in the end of the ex vivo stimulation of the colonic biopsies. | Immune system reinforcement will be evaluated after 90 minutes of ex vivo stimulation of the colonic biopsies.
  Selected pro- and anti- inflammatory cytokines levels will be measured on the colonic biopsies tissues by ELISA techniques.
Gastrointestinal health status prior to the initiation of the study. | Gastrointestinal health will be measured at baseline prior to the initiation of the study as background information.
  Gastrointestinal health will be evaluated once with the use of a 1-day questionnaire consisting of 13 items concerning satiety, abdominal pain, diarrhoea, constipation and bloating.The intensity of each parameter will be assessed on a scale of 0-7, where '0' represents absence of symptoms and '7' severe symptoms.
Dietary intake prior to the initiation of the study. | Dietary intake will be measured at baseline prior to the initiation of the study as background information.
  Dietary intake will be evaluated with the use of 3-days diet intake records.
Dietary habits prior to the initiation of the study. | Dietary habits will be measured at baseline prior to the initiation of the study as background information.
  Dietary habits will be evaluated with the use of food frequency questionnaire (FFQ).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brummer, Professor, Principal Investigator — Örebro University, School of Medical Sciences, Sweden
Locations (1):
- Campus USÖ, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Research center website — https://www.oru.se/english/research/research-environments/mh/nutrition-gut-brain-interactions-research-centre-ngbi/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT05421793/Prot_SAP_000.pdf